CLINICAL TRIAL: NCT00179608
Title: Phase I Safety Study of the Combination of Lenalidomide and DTIC (Dacarbazine) in Patients With Metastatic Malignant Melanoma Previously Untreated With Systemic Chemotherapy
Brief Title: Study of the Combination of Lenalidomide and DTIC (Dacarbazine) in Patients With Metastatic Malignant Melanoma Previously Untreated With Systemic Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Prologue Research International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MEL-003
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Malignant Melanoma
Keywords: CC-5013; CC5013; celgene; Melanoma; Revlimid; Metastatic Malignant Melanoma; Lenalidomide
MeSH Terms: conditions — Melanoma | interventions — Lenalidomide

INTERVENTIONS:
Drug: CC-5013

SUMMARY:
This study will determine the MDT of intravenous DTIC when administered in combination with a fixed dose of oral lenalidomide in subjects with metastatic malignant melanoma previously untreated with systemic chemotherapy. This study will evaluate the safety and preliminary efficacy of the combination of lenalidomide and DTIC. Subjects will be receive lenalidomide for 14 consecutive days and DTIC on day one of each 21 day cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document
2. Age greater than or equal to 18 years at the time of signing Informed Consent
3. Be able to adhere to the study visit schedule and other protocol requirements
4. Histological documentation of malignant melanoma with evidence of metastatic disease
5. For the 10 patients enrolled at the MTD, at least one measurable lesion must be present (see Appendix II)
6. ECOG performance status of 0, 1 or 2 (see Appendix I)
7. Laboratory tests within these ranges:

   1. Absolute neutrophil count greater than or equal to 1,500/uL
   2. Platelet count greater than or equal to 100,000/uL
   3. Serum creatinine less than or equal to 1.5 mg/dL
   4. Total bilirubin less that or equal to 1.5 mg.dL
   5. AST (SGOT) / ALT (SGPT) less than or equal to to 2 times upper limit of normal (ULN)
8. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug.

   In addition, sexually active WCBP must agree to use at least two methods of adequate contraceptive (oral, injectable, or implantable hormonal contraceptive, tubal ligation, intra-uterine device, barrier contraceptive with spermicide, contraceptive skin patch or vasectomized partner) while on study drug
9. All acute adverse effects (excluding alopecia of any prior therapy must have resolved to less than or equal to grade 1 (NCI CTCAE v3.0)
10. Patients must be able to take medications orally

Exclusion Criteria:

1. Pregnant or lactating females
2. Any serious medical condition, including psychiatric illnesses that will prevent the patient from signing the informed consent or place the patient at an unacceptable risk if he/she participates in the study.
3. Prior treatment with systemic chemotherapy. Patients who have received prior immunotherapy, including thalidomide, or radiotherapy remain eligible.

   Lesions within a prior field of radiation may only be used as indicator lesions if there has been evidence of disease progression at that site.
4. Prior history of malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the patient has been free of the disease for at least 3 years.
5. Use of thalidomide or biologic response modifier therapy within 14 days of Day 1, Cycle 1
6. Prior greater than or equal to grade 2 allergic reaction to thalidomide
7. Prior desquamating rash while taking thalidomide
8. Any prior use of lenalidomide
9. Concurrent use of any other anti-cancer agents
10. Radiation or surgical treatment of melanoma within 28 days of starting study treatment
11. Active infection
12. Central nervous system (CNS) metastases
13. Patients with > grade-2 neuropathy
14. Patients with known HIV positivity or AIDS-related illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2005-09-01 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2007-06-01 (Actual)

PRIMARY OUTCOMES:
To determine MTD of intravenous DTIC during the first 2 cycles (6 wks) of treatment

SECONDARY OUTCOMES:
To evaluate the safety profile of combination lenalidomide plus DTIC, the preliminary efficacy of combination lenalidomide plus DTIC
To define the recommended phase II doses of lenalidomide and DTIC when administered as combination therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Hwu WJ, Knight RD, Patnana M, Bassett R, Papadopoulos NE, Kim KB, Hwu P, Bedikian A. Phase I safety study of lenalidomide and dacarbazine in patients with metastatic melanoma previously untreated with systemic chemotherapy. Melanoma Res. 2010 Dec;20(6):501-6. doi: 10.1097/CMR.0b013e32833faf18. PMID 20859231